CLINICAL TRIAL: NCT06513026
Title: Milk for Diabetes Prevention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Dairy Council (Other); University of Minnesota (UM) Advanced Research and Diagnostic Laboratory (ARDL) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-16045
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Lactose Intolerance; Lactose Intolerant; Lactase Persistence; Pre-Diabetes; Diabetes Mellitus, Type 2
Keywords: Lactose; Lactose-free; Lactase Non Persistence
MeSH Terms: conditions — Lactose Intolerance; Glucose Intolerance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactose-Containing Milk (Active Comparator): Participants will be randomized to lactose-containing milk in strata of age (<60, ≥60) and sex (female, male). Within each age and sex stratum, 10 participants will be randomized into two intervention groups in a 1:1 ratio
  Interventions: Dietary Supplement: Lactose-Containing Milk
- Lactose-Free Milk (Active Comparator): Participants will be randomized to lactose-free milk in strata of age (<60, ≥60) and sex (female, male). Within each age and sex stratum, 10 participants will be randomized into two intervention groups in a 1:1 ratio
  Interventions: Dietary Supplement: Lactose-Free Milk

INTERVENTIONS:
Dietary Supplement: Lactose-Containing Milk — Participants will be asked to drink regular milk (1% or 2%) for 12 weeks as follows:
  * Weeks 1-4: ½ cup milk per day
  * Weeks 5-8: 1 cup milk per day
  * Weeks 9-12: 2 cups milk per day
  Participants will continue drinking 2 cups milk/day for 2 weeks after the 12-week follow-up visit.
  Arms: Lactose-Containing Milk
Dietary Supplement: Lactose-Free Milk — Participants will be asked to drink 1% or 2% lactose-free milk for 12 weeks as follows:
  * Weeks 1-4: ½ cup milk per day
  * Weeks 5-8: 1 cup milk per day
  * Weeks 9-12: 2 cups milk per day
  Participants will continue drinking 2 cups milk/day for 2 weeks after the 12-week follow-up visit.
  Arms: Lactose-Free Milk

SUMMARY:
Individuals with lactase non-persistence (LNP; determined by a functional variant in the LCT gene [rs4988235, GG genotype]) are susceptible to lactose intolerance in adulthood due to deficiency of lactase, the enzyme which digests milk lactose sugars. However, many LNP individuals still drink ≥1 cup of milk daily. Recent analysis in the Hispanic Community Health Study/Study of Latinos (HCHS/SOL) found that consumption of 1 serving (cup) of milk/day was associated with ~30% lower risk of type 2 diabetes among LNP individuals, but not among individuals with lactase persistence (LP). This beneficial effect might be partially explained by favorable alterations in gut microbiota and related metabolites associated with higher milk consumption among LNP individuals. Based on these observational study findings, the investigator team proposes to conduct a randomized, controlled trial of lactose-containing vs. lactose-free milk in LNP individuals with pre-diabetes, to comprehensively investigate the effects of milk intake on the gut microbiome and glycemic outcomes.

DETAILED DESCRIPTION:
The trial will feature a 2-week milk washout period, followed by 1:1 randomization to lactose-containing (1% or 2%) or lactose-free (1% or 2%) milk for 12 weeks (4 weeks each of ½ cup, 1 cup, and 2 cups milk). Before and after the 12 weeks, visits will entail lactose challenge hydrogen breath tests (HBT; i.e., lactose tolerance tests) and blood tests for fasting glucose, hemoglobin A1c, and metabolomics; while stool samples and continuous glucose monitoring (CGM) data will be collected at home using provided kits/devices.

Specific aims of the study are to: (1) establish feasibility and tolerability of a randomized trial of lactose-containing vs. lactose-free milk; (2) to examine the effect of lactose-containing milk on gut microbiome species, functions, and metabolites in LNP individuals with pre-diabetes; and (3) to examine the effect of lactose-containing milk on glycemic outcomes in LNP individuals with pre-diabetes.

ELIGIBILITY:
Inclusion Criteria:

* LNP genotype (LCT gene rs4988235, GG genotype)
* History of pre-diabetes, defined as fasting blood glucose 100-125 mg/dL and/or hemoglobin A1c (HbA1c) 5.7-6.4% and have not been diagnosed with diabetes nor take diabetes medication (pre-diabetes determined at most recent study visit [for HCHS/SOL participant] or most recent medical chart or self-report [for other participant])
* Drink ≤1 cup milk/day
* Basic computer or smartphone skills
* Can speak and read English fluently

Exclusion Criteria:

* Diabetes diagnosis
* Taking anti-diabetes medication
* Cancer, cardiovascular disease (CVD), or life-threatening illness
* Known milk allergy
* Has severe GI symptoms after drinking milk
* History of GI surgery
* Had a double mastectomy
* Smoking
* More than 1 alcoholic beverage/day
* Pregnant or breastfeeding
* Colonoscopy in last 2 weeks
* Antibiotics in last 3 months
* Taking probiotics or fiber supplements (if taking, must be able to stop taking during study)
* Taking laxatives, stool softeners, anti-diarrheal (if taking, must be able to stop taking during study)
* Taking lactase pills (if taking, must be able to stop taking)
* Participating in extreme dieting program
* Planning extended travel that would prevent participation in study
* Taking medication that must be taken separate from calcium or dairy products

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Stratified in a 1:1 ratio
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal symptoms | Daily From Screening visit to Week 12
  Gastrointestinal symptoms, specifically abdominal pain, bloating, flatulence, and diarrhea, will be recorded daily from screening visit through 12 weeks of milk intervention. The occurrence and severity of these four adverse events will be summarized and reported by study arm. Average frequencies of none-mild vs. moderate-severe symptoms will be compared between treatment groups by week of study, as well as for specific time intervals corresponding to milk doses (weeks 1-4, 5-8, 9-12).
Change in Expired Breath Hydrogen | From Baseline to Week 12
  Expired breath hydrogen after lactose challenge will be measured during the baseline visit and after 12 weeks of milk intervention at the time of the follow-up visit using Hydrogen Breath Test (HBT) kits. Breath tubes will be mailed to an external laboratory where stable isotope analysis for expired breath hydrogen will be conducted. Expired breath hydrogen will be expressed as incremental Area Under the Curve (iAUC). Change in iAUC from baseline to week 12 will be summarized using basic descriptive statistics (group means and standard deviations), and change in iAUC will be compared between treatment groups.
Change in gut microbiome features - Relative Abundance of Species | From Baseline to Week 12
  Stool samples will be collected using home stool microbiome kits at baseline, 4-, 8-, and 12-week timepoints. Shotgun sequencing will be conducted. Change in relative abundance of species (with >1% mean relative abundance) from baseline will summarized, using basic descriptive statistics (group means and standard deviations). Change in relative abundance of species from baseline will be compared between the treatment groups.
Change in gut microbiome features - Functional Pathway Relative Abundance | From Baseline to Week 12
  Stool samples will be collected using home stool microbiome kits at baseline, 4-, 8-, and 12-week timepoints. Shotgun sequencing will be conducted. Change in relative abundance of functional pathways (with >1% mean relative abundance) from baseline will summarized, using basic descriptive statistics (group means and standard deviations). Change in relative abundance of functional pathways from baseline will be compared between the treatment groups.
Change in gut microbiome features - Metabolomics | From Baseline to Week 12
  Targeted metabolic profiling will be performed on serum and stool samples (baseline and week 12) using LC-MS/MS methods for absolute quantitation of 70 metabolites associated with gut bacterial metabolism. Change in stool and serum metabolites from baseline will be summarized using basic descriptive statistics (group means and standard deviations). Change in stool and serum metabolites from baseline will be compared between the treatment groups.
Change in glycemic outcomes - Fasting glucose | From Baseline to Week 12
  Blood sera samples for fasting glucose will be collected at baseline and Week 12. Fasting glucose, i.e., blood sugar levels following an 8-hour fast, will be analyzed via standard analytical chemistry approaches and reported in mg/dL or mmol/L units. Ranges vary but a fasting glucose level <99 mg/dL is considered 'normal', between 100-125 mg/dL is within the 'pre-diabetic' range, >126 mg/dL is within the 'diabetic' range. Change in fasting glucose from baseline will be summarized using descriptive statistics (means and standard deviations) and compared between the treatment groups.
Change in glycemic outcomes - Hemoglobin A1c (HbA1c) | From Baseline to Week 12
  Whole blood samples for HbA1c will be collected at baseline and Week 12. HbA1c, used to measure the amount of hemoglobin with attached glucose and reflects average blood glucose levels over the past several months, will be analyzed via standard analytical chemistry approaches. Ranges vary, however, a 'normal' HbA1c is generally <5.7%, 5.7-6.4% is in the 'pre-diabetic' range and a value of 6.5% or greater is in the 'diabetic' range. Change in HbA1c from baseline will be summarized using descriptive statistics (means and standard deviations) and compared between the treatment groups.
Change in glycemic outcomes - Continuous Glucose Monitoring (CGM) mean glucose | From Screening visit to Week 14 visit
  During screening visit participants will have a 2-week continuous glucose monitor (CGM) applied to the skin on the upper arm in advance of the 2-week milk washout period. The CGM will be returned during the baseline visit 2 weeks later. After the 12 week visit, another 2-week CGM will be applied during which time participants will continue drinking milk concurrent with the 2-week CGM (i.e., until 14 weeks). Change in mean glucose (mg/dL) from screening to week 14 will be summarized using descriptive statistics (means and standard deviations) and compared between the treatment groups.
Change in glycemic outcomes - Continuous Glucose Monitoring (CGM) glycemic variability | From Screening visit to Week 14 visit
  During screening visit participants will have a 2-week continuous glucose monitor (CGM) applied to the skin on the upper arm in advance of the 2-week milk washout period. The CGM will be returned during the baseline visit 2 weeks later. After the 12 week visit, another 2-week CGM will be applied during which time participants will continue drinking milk concurrent with the 2-week CGM (i.e., until 14 weeks). Change in glycemic variability (%CV) from screening to week 14 will be summarized using descriptive statistics (means and standard deviations) and compared between the treatment groups.
Change in glycemic outcomes - Continuous Glucose Monitoring (CGM) time above range | From Screening visit to Week 14 visit
  During screening visit participants will have a 2-week continuous glucose monitor (CGM) applied to the skin on the upper arm in advance of the 2-week milk washout period. The CGM will be returned during the baseline visit 2 weeks later. After the 12 week visit, another 2-week CGM will be applied during which time participants will continue drinking milk concurrent with the 2-week CGM (i.e., until 14 weeks). Change in time above range (%) from screening to week 14 will be summarized using descriptive statistics (means and standard deviations) and compared between the treatment groups.
Change in glycemic outcomes - Continuous Glucose Monitoring (CGM) time in range | From Screening visit to Week 14 visit
  During screening visit participants will have a 2-week continuous glucose monitor (CGM) applied to the skin on the upper arm in advance of the 2-week milk washout period. The CGM will be returned during the baseline visit 2 weeks later. After the 12 week visit, another 2-week CGM will be applied during which time participants will continue drinking milk concurrent with the 2-week CGM (i.e., until 14 weeks). Change in time in range (%) from screening to week 14 will be summarized using descriptive statistics (means and standard deviations) and compared between the treatment groups.
Change in glycemic outcomes - Continuous Glucose Monitoring (CGM) time below range | From Screening visit to Week 14 visit
  During screening visit participants will have a 2-week continuous glucose monitor (CGM) applied to the skin on the upper arm in advance of the 2-week milk washout period. The CGM will be returned during the baseline visit 2 weeks later. After the 12 week visit, another 2-week CGM will be applied during which time participants will continue drinking milk concurrent with the 2-week CGM (i.e., until 14 weeks). Change in time below range (%) from screening to week 14 will be summarized using descriptive statistics (means and standard deviations) and compared between the treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Brandilyn Peters-Samuelson, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- HCHS/SOL Bronx Field Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Background] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Background] Parker ED, Lin J, Mahoney T, Ume N, Yang G, Gabbay RA, ElSayed NA, Bannuru RR. Economic Costs of Diabetes in the U.S. in 2022. Diabetes Care. 2024 Jan 1;47(1):26-43. doi: 10.2337/dci23-0085. PMID 37909353
- [Background] Uusitupa M, Khan TA, Viguiliouk E, Kahleova H, Rivellese AA, Hermansen K, Pfeiffer A, Thanopoulou A, Salas-Salvado J, Schwab U, Sievenpiper JL. Prevention of Type 2 Diabetes by Lifestyle Changes: A Systematic Review and Meta-Analysis. Nutrients. 2019 Nov 1;11(11):2611. doi: 10.3390/nu11112611. PMID 31683759
- [Background] Wareham NJ. Personalised prevention of type 2 diabetes. Diabetologia. 2022 Nov;65(11):1796-1803. doi: 10.1007/s00125-022-05774-7. Epub 2022 Aug 2. PMID 35916901
- [Background] Liu B, Sun Y, Bao W. Creating and supporting a healthy food environment for type 2 diabetes prevention. Lancet Planet Health. 2018 Oct;2(10):e423-e424. doi: 10.1016/S2542-5196(18)30211-0. No abstract available. PMID 30318098
- [Background] Aune D, Norat T, Romundstad P, Vatten LJ. Dairy products and the risk of type 2 diabetes: a systematic review and dose-response meta-analysis of cohort studies. Am J Clin Nutr. 2013 Oct;98(4):1066-83. doi: 10.3945/ajcn.113.059030. Epub 2013 Aug 14. PMID 23945722
- [Background] Luo K, Chen GC, Zhang Y, Moon JY, Xing J, Peters BA, Usyk M, Wang Z, Hu G, Li J, Selvin E, Rebholz CM, Wang T, Isasi CR, Yu B, Knight R, Boerwinkle E, Burk RD, Kaplan RC, Qi Q. Variant of the lactase LCT gene explains association between milk intake and incident type 2 diabetes. Nat Metab. 2024 Jan;6(1):169-186. doi: 10.1038/s42255-023-00961-1. Epub 2024 Jan 22. PMID 38253929
- [Background] Segurel L, Bon C. On the Evolution of Lactase Persistence in Humans. Annu Rev Genomics Hum Genet. 2017 Aug 31;18:297-319. doi: 10.1146/annurev-genom-091416-035340. Epub 2017 Apr 19. PMID 28426286
- [Background] Storhaug CL, Fosse SK, Fadnes LT. Country, regional, and global estimates for lactose malabsorption in adults: a systematic review and meta-analysis. Lancet Gastroenterol Hepatol. 2017 Oct;2(10):738-746. doi: 10.1016/S2468-1253(17)30154-1. Epub 2017 Jul 7. PMID 28690131
- [Background] Anguita-Ruiz A, Aguilera CM, Gil A. Genetics of Lactose Intolerance: An Updated Review and Online Interactive World Maps of Phenotype and Genotype Frequencies. Nutrients. 2020 Sep 3;12(9):2689. doi: 10.3390/nu12092689. PMID 32899182
- [Background] Robles L, Priefer R. Lactose Intolerance: What Your Breath Can Tell You. Diagnostics (Basel). 2020 Jun 17;10(6):412. doi: 10.3390/diagnostics10060412. PMID 32560312
- [Background] Wilt TJ, Shaukat A, Shamliyan T, Taylor BC, MacDonald R, Tacklind J, Rutks I, Schwarzenberg SJ, Kane RL, Levitt M. Lactose intolerance and health. Evid Rep Technol Assess (Full Rep). 2010 Feb;(192):1-410. PMID 20629478
- [Background] JanssenDuijghuijsen L, Looijesteijn E, van den Belt M, Gerhard B, Ziegler M, Ariens R, Tjoelker R, Geurts J. Changes in gut microbiota and lactose intolerance symptoms before and after daily lactose supplementation in individuals with the lactase nonpersistent genotype. Am J Clin Nutr. 2024 Mar;119(3):702-710. doi: 10.1016/j.ajcnut.2023.12.016. Epub 2023 Dec 28. PMID 38159728
- [Background] Carroccio A, Montalto G, Cavera G, Notarbatolo A. Lactose intolerance and self-reported milk intolerance: relationship with lactose maldigestion and nutrient intake. Lactase Deficiency Study Group. J Am Coll Nutr. 1998 Dec;17(6):631-6. doi: 10.1080/07315724.1998.10718813. PMID 9853544
- [Background] Zheng X, Chu H, Cong Y, Deng Y, Long Y, Zhu Y, Pohl D, Fried M, Dai N, Fox M. Self-reported lactose intolerance in clinic patients with functional gastrointestinal symptoms: prevalence, risk factors, and impact on food choices. Neurogastroenterol Motil. 2015 Aug;27(8):1138-46. doi: 10.1111/nmo.12602. Epub 2015 Jun 19. PMID 26095206
- [Background] Agus A, Planchais J, Sokol H. Gut Microbiota Regulation of Tryptophan Metabolism in Health and Disease. Cell Host Microbe. 2018 Jun 13;23(6):716-724. doi: 10.1016/j.chom.2018.05.003. PMID 29902437
- [Background] Qi Q, Li J, Yu B, Moon JY, Chai JC, Merino J, Hu J, Ruiz-Canela M, Rebholz C, Wang Z, Usyk M, Chen GC, Porneala BC, Wang W, Nguyen NQ, Feofanova EV, Grove ML, Wang TJ, Gerszten RE, Dupuis J, Salas-Salvado J, Bao W, Perkins DL, Daviglus ML, Thyagarajan B, Cai J, Wang T, Manson JE, Martinez-Gonzalez MA, Selvin E, Rexrode KM, Clish CB, Hu FB, Meigs JB, Knight R, Burk RD, Boerwinkle E, Kaplan RC. Host and gut microbial tryptophan metabolism and type 2 diabetes: an integrative analysis of host genetics, diet, gut microbiome and circulating metabolites in cohort studies. Gut. 2022 Jun;71(6):1095-1105. doi: 10.1136/gutjnl-2021-324053. Epub 2021 Jun 14. PMID 34127525
- [Background] Gojda J, Cahova M. Gut Microbiota as the Link between Elevated BCAA Serum Levels and Insulin Resistance. Biomolecules. 2021 Sep 28;11(10):1414. doi: 10.3390/biom11101414. PMID 34680047
- [Background] Guha S, Majumder K. Comprehensive Review of gamma-Glutamyl Peptides (gamma-GPs) and Their Effect on Inflammation Concerning Cardiovascular Health. J Agric Food Chem. 2022 Jul 6;70(26):7851-7870. doi: 10.1021/acs.jafc.2c01712. Epub 2022 Jun 21. PMID 35727887
- [Background] Li X, Yin J, Zhu Y, Wang X, Hu X, Bao W, Huang Y, Chen L, Chen S, Yang W, Shan Z, Liu L. Effects of Whole Milk Supplementation on Gut Microbiota and Cardiometabolic Biomarkers in Subjects with and without Lactose Malabsorption. Nutrients. 2018 Oct 2;10(10):1403. doi: 10.3390/nu10101403. PMID 30279333
- [Background] Aguayo-Mazzucato C, Diaque P, Hernandez S, Rosas S, Kostic A, Caballero AE. Understanding the growing epidemic of type 2 diabetes in the Hispanic population living in the United States. Diabetes Metab Res Rev. 2019 Feb;35(2):e3097. doi: 10.1002/dmrr.3097. Epub 2018 Dec 4. PMID 30445663
- [Background] Ugidos-Rodriguez S , Matallana-Gonzalez MC , Sanchez-Mata MC . Lactose malabsorption and intolerance: a review. Food Funct. 2018 Aug 15;9(8):4056-4068. doi: 10.1039/c8fo00555a. PMID 29999504
- [Background] Kaplan RC, Wang Z, Usyk M, Sotres-Alvarez D, Daviglus ML, Schneiderman N, Talavera GA, Gellman MD, Thyagarajan B, Moon JY, Vazquez-Baeza Y, McDonald D, Williams-Nguyen JS, Wu MC, North KE, Shaffer J, Sollecito CC, Qi Q, Isasi CR, Wang T, Knight R, Burk RD. Gut microbiome composition in the Hispanic Community Health Study/Study of Latinos is shaped by geographic relocation, environmental factors, and obesity. Genome Biol. 2019 Nov 1;20(1):219. doi: 10.1186/s13059-019-1831-z. PMID 31672155
- [Background] Wang Z, Peters BA, Bryant M, Hanna DB, Schwartz T, Wang T, Sollecito CC, Usyk M, Grassi E, Wiek F, Peter LS, Post WS, Landay AL, Hodis HN, Weber KM, French A, Golub ET, Lazar J, Gustafson D, Sharma A, Anastos K, Clish CB, Burk RD, Kaplan RC, Knight R, Qi Q. Gut microbiota, circulating inflammatory markers and metabolites, and carotid artery atherosclerosis in HIV infection. Microbiome. 2023 May 27;11(1):119. doi: 10.1186/s40168-023-01566-2. PMID 37237391
- [Background] Sanders JG, Nurk S, Salido RA, Minich J, Xu ZZ, Zhu Q, Martino C, Fedarko M, Arthur TD, Chen F, Boland BS, Humphrey GC, Brennan C, Sanders K, Gaffney J, Jepsen K, Khosroheidari M, Green C, Liyanage M, Dang JW, Phelan VV, Quinn RA, Bankevich A, Chang JT, Rana TM, Conrad DJ, Sandborn WJ, Smarr L, Dorrestein PC, Pevzner PA, Knight R. Optimizing sequencing protocols for leaderboard metagenomics by combining long and short reads. Genome Biol. 2019 Oct 31;20(1):226. doi: 10.1186/s13059-019-1834-9. PMID 31672156
- [Background] Langmead B, Salzberg SL. Fast gapped-read alignment with Bowtie 2. Nat Methods. 2012 Mar 4;9(4):357-9. doi: 10.1038/nmeth.1923. PMID 22388286
- [Background] Zhu Q, Huang S, Gonzalez A, et al. OGUs enable effective, phylogeny-aware analysis of even shallow metagenome community structures. 2021:2021.04.04.438427. doi:10.1101/2021.04.04.438427 %J bioRxiv
- [Background] Kanehisa M, Sato Y, Kawashima M, Furumichi M, Tanabe M. KEGG as a reference resource for gene and protein annotation. Nucleic Acids Res. 2016 Jan 4;44(D1):D457-62. doi: 10.1093/nar/gkv1070. Epub 2015 Oct 17. PMID 26476454
- [Background] Caspi R, Billington R, Keseler IM, Kothari A, Krummenacker M, Midford PE, Ong WK, Paley S, Subhraveti P, Karp PD. The MetaCyc database of metabolic pathways and enzymes - a 2019 update. Nucleic Acids Res. 2020 Jan 8;48(D1):D445-D453. doi: 10.1093/nar/gkz862. PMID 31586394
- [Background] McMurdie PJ, Holmes S. phyloseq: an R package for reproducible interactive analysis and graphics of microbiome census data. PLoS One. 2013 Apr 22;8(4):e61217. doi: 10.1371/journal.pone.0061217. Print 2013. PMID 23630581
- [Background] Oksanen J, Blanchet FG, Kindt R, et al. Multivariate analysis of ecological communities in R: vegan tutorial. R package version 1.7. 01/01 2013;
- [Background] Chen J, Bittinger K, Charlson ES, Hoffmann C, Lewis J, Wu GD, Collman RG, Bushman FD, Li H. Associating microbiome composition with environmental covariates using generalized UniFrac distances. Bioinformatics. 2012 Aug 15;28(16):2106-13. doi: 10.1093/bioinformatics/bts342. Epub 2012 Jun 17. PMID 22711789
- [Background] Turner-McGrievy GM, Wirth MD, Shivappa N, Wingard EE, Fayad R, Wilcox S, Frongillo EA, Hebert JR. Randomization to plant-based dietary approaches leads to larger short-term improvements in Dietary Inflammatory Index scores and macronutrient intake compared with diets that contain meat. Nutr Res. 2015 Feb;35(2):97-106. doi: 10.1016/j.nutres.2014.11.007. Epub 2014 Dec 3. PMID 25532675
- [Background] Thompson FE, Dixit-Joshi S, Potischman N, Dodd KW, Kirkpatrick SI, Kushi LH, Alexander GL, Coleman LA, Zimmerman TP, Sundaram ME, Clancy HA, Groesbeck M, Douglass D, George SM, Schap TE, Subar AF. Comparison of Interviewer-Administered and Automated Self-Administered 24-Hour Dietary Recalls in 3 Diverse Integrated Health Systems. Am J Epidemiol. 2015 Jun 15;181(12):970-8. doi: 10.1093/aje/kwu467. Epub 2015 May 10. PMID 25964261
- [Background] Lavange LM, Kalsbeek WD, Sorlie PD, Aviles-Santa LM, Kaplan RC, Barnhart J, Liu K, Giachello A, Lee DJ, Ryan J, Criqui MH, Elder JP. Sample design and cohort selection in the Hispanic Community Health Study/Study of Latinos. Ann Epidemiol. 2010 Aug;20(8):642-9. doi: 10.1016/j.annepidem.2010.05.006. PMID 20609344
- [Background] Sorlie PD, Aviles-Santa LM, Wassertheil-Smoller S, Kaplan RC, Daviglus ML, Giachello AL, Schneiderman N, Raij L, Talavera G, Allison M, Lavange L, Chambless LE, Heiss G. Design and implementation of the Hispanic Community Health Study/Study of Latinos. Ann Epidemiol. 2010 Aug;20(8):629-41. doi: 10.1016/j.annepidem.2010.03.015. PMID 20609343
- [Background] Gloor GB, Macklaim JM, Pawlowsky-Glahn V, Egozcue JJ. Microbiome Datasets Are Compositional: And This Is Not Optional. Front Microbiol. 2017 Nov 15;8:2224. doi: 10.3389/fmicb.2017.02224. eCollection 2017. PMID 29187837
- See also: R: A language and environment for statistical computing. R Foundation for Statistical Computing; 2021. — https://www.r-project.org/